CLINICAL TRIAL: NCT05024786
Title: The Effect of Continuous Quality Improvement on the Outcome of Patients Supported With Extracorporeal Membrane Oxygenation in ICU
Brief Title: The Effect of CQI on the Outcome of Patients Supported With ECMO
Status: Completed | Type: Observational
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, JinyanXing, Director, The Affiliated Hospital of Qingdao University
Other Study IDs: QYFYKYLL931311921
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Respiratory and Circulation Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group
- CQI group
  Interventions: Other: continuous quality improvements

INTERVENTIONS:
Other: continuous quality improvements — We implement the continuous quality improvement strategy in CQI group, and observe the effect of the strategy on the mortality of patients supported with ECMO .
  Groups: CQI group

SUMMARY:
This was a prospective observational study in comparison with a retrospective control group(Jan 2015 to Jun 2019). Two ICUs in China were included. The continuous quality improvement (CQI)strategies were implemented from Jul 2019 to Jun 2021(CQI group). The mortalities of ECMO patients was compared between the CQI group and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old who received ECMO support in the centers

Exclusion Criteria:

* patients waiting for transplantation with ECMO.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old who received ECMO support in the centers between January 2015 and April 2021 were included, not including patients waiting for transplantation with ECMO.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
The mortality of patients supported with ECMO | January, 2021 to July, 2021

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jing Y, Yuan Z, Zhou W, Han X, Qi Q, Song K, Xing J. A phased intervention bundle to decrease the mortality of patients with extracorporeal membrane oxygenation in intensive care unit. Front Med (Lausanne). 2022 Oct 17;9:1005162. doi: 10.3389/fmed.2022.1005162. eCollection 2022. PMID 36325385